CLINICAL TRIAL: NCT00037453
Title: Analysis of Sex Hormones and Lipoproteins in Young Males
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1172; R03HL065728 (NIH)
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2004-08

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Heart Diseases
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Heart Diseases

SUMMARY:
To analyze the relationship of sex hormones to lipoproteins in young males.

DETAILED DESCRIPTION:
BACKGROUND:

The investigators conducted a secondary analysis of the Sex Hormones and Lipoproteins in Adolescent Males Study (HD/HL18281), a 3-year (1984-1987) study of lipids, blood pressure, weight, fat patterning, and sex steroid hormones (SSH) in adolescent males. A total of 664 black and white males, ages 10-15, were enrolled into a study designed as a series of repeated data collections over two years within age cohorts. Cross-sectional analyses were used to explain differences during adolescence in sex steroid hormones and sex steroid hormone-lipid relationships between black and white boys and between boys with and without a family history of coronary heart disease.. When the data were originally collected for this study, theoretical models of flexible longitudinal analytic techniques had been developed, but were not available for computer use. These techniques, now supported by software, allow a more powerful and complete analysis of these data.

DESIGN NARRATIVE:

The primary aim of these analyses was to explain the contribution of changes in sex steroid hormones and fat patterning to changes in plasma concentrations of high (HDL-C) and low (LDL-C) density lipoprotein cholesterol, triglycerides (TG), and apolipoproteins (apo) Al, All, and B occurring during puberty in males. Sex steroid hormones assayed included estradiol (E2) and free testosterone (T). The following hypotheses were tested: (1) increasing free T predicts/leads to decreases in HDL-C and increases in LDL-C, apo B, and the LDL-C/HDL-C ratio in adolescent males; (2) increasing E2 predicts decreases in apo B, LDL-C and the LDL-C/HDL- C ratio, but the resultant effects will vary with adiposity and fat patterning; (3) rapid weight gain predicts increased central adiposity, defined as the ratio of truncal skinfolds to total skinfolds, and with greater decreases in HDL-C and increases in triglycerides, apo B, LDL-C and the LDL- C/HDL-C ratio. Rapid weight gain predicts increased E2, but the atherogenic effects of increased central adiposity on lipids are greater than the anti- atherogenic effects of E2. These analyses provided a better understanding of metabolic factors underlying obesity-hormone-lipoprotein relationships.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Ages: 10 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2001-04; Study Completion 2003-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Barton — Maryland Medical Research Institute

REFERENCES:
- [Background] Morrison JA, Barton BA, Biro FM, Sprecher DL. Sex hormones and the changes in adolescent male lipids: longitudinal studies in a biracial cohort. J Pediatr. 2003 Jun;142(6):637-42. doi: 10.1067/mpd.2003.246. PMID 12838191